CLINICAL TRIAL: NCT05168527
Title: An Open Single-center Phase II Clinical Study of Fruquintinib Combined With Chemotherapy in Patients With Liver Metastases From Pancreatic Cancer
Brief Title: The First Line Treatment of Fruquintinib Combined With Albumin Paclitaxel and Gemcitabine in Pancreatic Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, President of Shanghai Pancreatic Cancer Institute, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-NG
Record Dates: First submitted 2021-12-08; First posted 2021-12-23 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Safety and Effectiveness; TKI; Chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): This is an opened single-arm phase 2 study， the study drug includes Fruquintinib combine with Paclitaxel Injection and Gemcitabine.
  Interventions: Drug: Fruquintinib,Albumin Paclitaxel,Gemcitabine

INTERVENTIONS:
Drug: Fruquintinib,Albumin Paclitaxel,Gemcitabine — The study will mainly explore the safety and tolerability of fixed-dose level of Fruquintinib (4 mg, continuous medication for 3 weeks and withdrawal for 1 week) combined with fixed-dose level of albumin paclitaxel and gemcitabine. The fixed dose of Fruquintinib is 4 mg, with a treatment cycle every 28 days. A 28-day observation window was used to explore the side effects of fruquintinib in the combined treatment of pancreatic cancer patients with liver metastases. Evaluable patients will be assessed for DLT within 28 days after the first administration of the study drug. The 24 patients enrolled in the follow-up group will mainly evaluate the initial efficacy of furquintinib combined with albumin paclitaxel and gemcitabine as the first-line standard treatment for patients with metastatic pancreatic cancer.

SUMMARY:
The aim of this study is to evaluate the safety and effectiveness of Fruquintinib combined with Albumin Paclitaxel and Gemcitabine on pancreatic cancer patients with liver metastases. Plan to enrollment 30 patients.

DETAILED DESCRIPTION:
Pancreatic cancer is the most deadly malignant tumor commonly found in the digestive system and is known as the king of cancer. According to the global cancer statistics released in 2018, there are about 458,900 new cases of pancreatic cancer worldwide each year, and the number of deaths due to pancreatic cancer each year is about 432,200. The data of pancreatic cancer collected by the National Cancer Center of China in 2019 showed that the incidence rate was 6.92 per 100,000, and new cases accounted for about 4.31% of all malignant tumors, ranking 10th; the case fatality rate was 6.16 per 100,000, with deaths every year It accounts for about 3.78% of all malignant tumors, ranking 7th. Compared with urban areas and rural areas, the morbidity and mortality have increased compared with previous years. The incidence of pancreatic cancer has been increasing year by year worldwide, and it is expected that by 2030, it will surpass colorectal cancer and breast cancer to become the second cancer-fatal tumor. Pancreatic cancer is extremely malignant, with a 5-year survival rate of only 9%, and its case fatality rate is basically equal to the incidence rate. The case fatality rate of pancreatic cancer may continue to rise, which will seriously threaten and affect human health.

The specific etiology and pathogenesis of pancreatic cancer are currently unclear, the early clinical manifestations are not obvious, the rapid development, the extremely high degree of malignancy, and the poor prognosis, all of which lead to the refractory and high mortality of pancreatic cancer. It is precisely because the early symptoms are not typical and the clinical signs are not obvious, most patients are already in the locally advanced stage or have distant metastases when they are diagnosed.In this case, the chance of surgical treatment is low and the effect is not ideal. 80% of pancreatic cancer patients are already in the inoperable advanced stage at the time of diagnosis, and more than 50% of them have found metastases at the time of diagnosis, and have lost the chance of radical surgery. The most common distant metastasis site is the liver. At present, for patients with liver metastases from pancreatic cancer, the standard treatment regimen in domestic and foreign guidelines is palliative treatment based on chemotherapy.

According to the latest updated treatment guidelines for metastatic pancreatic cancer by the American Society of Clinical Oncology (ASCO), the first-line chemotherapy regimen should be selected based on the patient's physical status. For patients with good physical status, a combination regimen may be considered, and patients with poor physical status should choose single-agent chemotherapy. Or the best supportive treatment. For those with good physical status, FOLFIRINOX, gemcitabine and paclitaxel are recommended; for patients with poor physical status, single-agent gemcitabine can be used. If tolerable, they can be combined with albumin paclitaxel or calciner under the guidance of an experienced oncologist. Petabine or erlotinib. Overall, the median OS of first-line chemotherapy did not exceed 12 months, and the median OS of second-line chemotherapy ranged from 3.3 to 9.9 months. Therefore, the overall treatment effect of pancreatic cancer was poor, and the median survival was only 6 months. For 8 months, the effect was not good. All major guidelines recommend the development of multi-center clinical studies to prolong patient survival and discover new effective drugs. In summary, actively exploring new comprehensive treatment strategies, breaking through treatment options for advanced pancreatic cancer, improving the survival time of patients with liver metastases of pancreatic cancer, and exploring the biological characteristics of liver metastases of pancreatic cancer are important clinical issues that urgently need to be resolved.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old;
2. Pancreatic cancer was confirmed by pathology or cytology;
3. Liver-metastatic confirmed by pathology or clinical imaging;
4. Newly treated patients who have not received any systemic treatment for pancreatic cancer are allowed to enter the group for patients who have previously used fluorouracils (excluding gemcitabine and or taxanes) as adjuvant treatments for recurrence;
5. ECOG score of preoperative physical condition was 0-1;
6. Expected survival time ≥3months;
7. There is at least one measurable lesion under CT evaluation according to the RECIST 1.1 standard,;
8. The patient has sufficient hematological function (not receiving blood, platelet transfusion or growth factor supportive therapy within 14 days before the start of the study treatment), determined according to the following laboratory test values:

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L;
   2. Platelets ≥ 100 × 109/L;
   3. Hemoglobin ≥ 9.0 g/dL;
9. The patient has sufficient liver and kidney function, which is determined according to the following laboratory test values:

   1. Serum creatinine ≤ 1.5 × ULN;
   2. If serum creatinine>1.5 × ULN, creatinine clearance rate ≥50ml/min;
   3. Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) in non-liver metastatic lesions ≤ 2.5 × ULN, and AST and ALT ≤ 5.0 × ULN in liver metastatic lesions;
   4. Serum albumin ≥ 2.5 g/dL;
   5. Total bilirubin ≤1.5 × ULN;
10. Men, women of childbearing age (postmenopausal women who must have been menopausal for at least 12 months to be considered infertile) and their partners voluntarily take it during treatment and at least six months after the last study drug is taken by the investigator. Effective contraceptive measures;
11. Able to understand and voluntarily sign a written informed consent form and voluntarily complete the research procedures and follow-up inspections. The informed consent form must be signed before the implementation of any research procedures specified by the trial

Exclusion Criteria:

1. Received chemotherapy within 14 days before entering the study.
2. Received VEGFR signaling pathway therapy or other anti-cancer therapy within 14 days before enrollment.
3. Received radiotherapy within 14 days before enrollment, and received chest radiotherapy within 28 days before enrollment.
4. Active central nervous system involvement is known.
5. Oral anticoagulant is being used, or an inhibitor or inducer of potent cytochrome oxidase 3A4 (CYP3A4) is being used (see Appendix 1 for details). Allow the use of subcutaneous anticoagulants.
6. Patients who have participated in clinical trials of reagents or new drugs under investigation within 28 days before the first treatment administration (phase I-IV clinical trials).
7. Adverse reactions caused by previous anti-tumor treatments did not recover to grade 1 or below (hair loss and peripheral neuropathy did not recover to grade 2 or below).
8. Active infection or unexplained fever> 38.5°C occurred within 2 weeks before the first administration (according to the judgment of the investigator, the subject can be included in the group for fever caused by the tumor).
9. Various chronic active infections, such as hepatitis B virus (evidence of hepatitis activity such as HBV-DNA ≥104 copies/ml or 2000IU/ml), hepatitis C and HIV.
10. Patients with elevated serum troponin T or I (above the normal limit specified by the research center).
11. Pregnant or lactating (lactating) women, where pregnancy is defined as the state of a woman after conception until the end of pregnancy, and the result of a serum β-human chorionic gonadotropin (β-hCG) laboratory test is confirmed to be positive.
12. Any of the following cardiac standards: the average QTcF calculated according to Fridericia's formula during the rest period of the screening period [QTcF = QT/(RR1/3), RR is the standardized heart rate value, obtained by dividing 60 by the heart rate]: male> 450 milliseconds , Female> 470 milliseconds; any clinically important abnormalities in the rhythm, conduction or morphology of the resting electrocardiogram (ECG) (for example, complete left bundle branch block, third degree heart block, second degree heart block); Congenital long QT syndrome or family history of long QT syndrome.
13. According to the investigator's judgment, patients who have not fully recovered after surgery, patients whose wounds are in an active healing stage, patients who underwent major surgery within 28 days before the start of the study, and patients who underwent minor surgery within 14 days before the start of the study.
14. Severe and uncontrollable accompanying diseases that may affect protocol compliance or interfere with the interpretation of results, including active opportunistic infections or advanced (severe) infections, and diabetes that cannot be controlled after adequate clinical anti-hyperglycemia treatment according to guidelines , Uncontrollable hypertension, cardiovascular disease (Class III or IV heart failure as defined by the New York Heart Association classification, heart block above II, congestive heart failure (CHF), myocardial infarction in the past 6 months , Unstable arrhythmia or unstable angina, cerebral infarction within 3 months, etc.) or lung disease (history of interstitial pneumonia, obstructive lung disease and symptomatic bronchospasm).
15. Any other situation that the researcher considers inappropriate to participate in clinical research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-03-02 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
ORR | through study completion, an average of 1 year
  Objective Response Rate

SECONDARY OUTCOMES:
PFS | through study completion, an average of 1 year
  Progression-free survival
DCR | through study completion, an average of 1 year
  Disease control Rate
OS | through study completion, an average of 1 year
  Overall Survival
DOR | through study completion, an average of 1 year
  Duration of Remission

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun MD Yu, PhD, Principal Investigator — Fudan University
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarez R, Musteanu M, Garcia-Garcia E, Lopez-Casas PP, Megias D, Guerra C, Munoz M, Quijano Y, Cubillo A, Rodriguez-Pascual J, Plaza C, de Vicente E, Prados S, Tabernero S, Barbacid M, Lopez-Rios F, Hidalgo M. Stromal disrupting effects of nab-paclitaxel in pancreatic cancer. Br J Cancer. 2013 Aug 20;109(4):926-33. doi: 10.1038/bjc.2013.415. Epub 2013 Aug 1. PMID 23907428
- [Background] Sankaranarayanan R. Cancer survival in Africa, Asia, the Caribbean and Central America. Introduction. IARC Sci Publ. 2011;(162):1-5. PMID 21675400
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Chiorean EG, Von Hoff DD, Reni M, Arena FP, Infante JR, Bathini VG, Wood TE, Mainwaring PN, Muldoon RT, Clingan PR, Kunzmann V, Ramanathan RK, Tabernero J, Goldstein D, McGovern D, Lu B, Ko A. CA19-9 decrease at 8 weeks as a predictor of overall survival in a randomized phase III trial (MPACT) of weekly nab-paclitaxel plus gemcitabine versus gemcitabine alone in patients with metastatic pancreatic cancer. Ann Oncol. 2016 Apr;27(4):654-60. doi: 10.1093/annonc/mdw006. Epub 2016 Jan 22. PMID 26802160
- [Background] Chu GC, Kimmelman AC, Hezel AF, DePinho RA. Stromal biology of pancreatic cancer. J Cell Biochem. 2007 Jul 1;101(4):887-907. doi: 10.1002/jcb.21209. PMID 17266048
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] da Rocha Lino A, Abrahao CM, Brandao RM, Gomes JR, Ferrian AM, Machado MC, Buzaid AC, Maluf FC, Peixoto RD. Role of gemcitabine as second-line therapy after progression on FOLFIRINOX in advanced pancreatic cancer: a retrospective analysis. J Gastrointest Oncol. 2015 Oct;6(5):511-5. doi: 10.3978/j.issn.2078-6891.2015.041. PMID 26487945
- [Background] Portal A, Pernot S, Tougeron D, Arbaud C, Bidault AT, de la Fouchardiere C, Hammel P, Lecomte T, Dreanic J, Coriat R, Bachet JB, Dubreuil O, Marthey L, Dahan L, Tchoundjeu B, Locher C, Lepere C, Bonnetain F, Taieb J. Nab-paclitaxel plus gemcitabine for metastatic pancreatic adenocarcinoma after Folfirinox failure: an AGEO prospective multicentre cohort. Br J Cancer. 2015 Sep 29;113(7):989-95. doi: 10.1038/bjc.2015.328. Epub 2015 Sep 15. PMID 26372701
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Eltawil KM, Renfrew PD, Molinari M. Meta-analysis of phase III randomized trials of molecular targeted therapies for advanced pancreatic cancer. HPB (Oxford). 2012 Apr;14(4):260-8. doi: 10.1111/j.1477-2574.2012.00441.x. Epub 2012 Feb 26. PMID 22404265
- [Background] Gilabert M, Chanez B, Rho YS, Giovanini M, Turrini O, Batist G, Kavan P, Raoul JL. Evaluation of gemcitabine efficacy after the FOLFIRINOX regimen in patients with advanced pancreatic adenocarcinoma. Medicine (Baltimore). 2017 Apr;96(16):e6544. doi: 10.1097/MD.0000000000006544. PMID 28422841
- [Background] Gill S, Ko YJ, Cripps C, Beaudoin A, Dhesy-Thind S, Zulfiqar M, Zalewski P, Do T, Cano P, Lam WYH, Dowden S, Grassin H, Stewart J, Moore M. PANCREOX: A Randomized Phase III Study of Fluorouracil/Leucovorin With or Without Oxaliplatin for Second-Line Advanced Pancreatic Cancer in Patients Who Have Received Gemcitabine-Based Chemotherapy. J Clin Oncol. 2016 Nov 10;34(32):3914-3920. doi: 10.1200/JCO.2016.68.5776. Epub 2016 Sep 30. PMID 27621395
- [Background] Hanahan D, Weinberg RA. The hallmarks of cancer. Cell. 2000 Jan 7;100(1):57-70. doi: 10.1016/s0092-8674(00)81683-9. No abstract available. PMID 10647931
- [Background] Hidalgo M. Pancreatic cancer. N Engl J Med. 2010 Apr 29;362(17):1605-17. doi: 10.1056/NEJMra0901557. No abstract available. PMID 20427809
- [Background] Hu J, Zhao G, Wang HX, Tang L, Xu YC, Ma Y, Zhang FC. A meta-analysis of gemcitabine containing chemotherapy for locally advanced and metastatic pancreatic adenocarcinoma. J Hematol Oncol. 2011 Mar 26;4:11. doi: 10.1186/1756-8722-4-11. PMID 21439076
- [Background] Ji Y, Liu P, Li Y, Bekele BN. A modified toxicity probability interval method for dose-finding trials. Clin Trials. 2010 Dec;7(6):653-63. doi: 10.1177/1740774510382799. Epub 2010 Oct 8. PMID 20935021
- [Background] Jones S, Zhang X, Parsons DW, Lin JC, Leary RJ, Angenendt P, Mankoo P, Carter H, Kamiyama H, Jimeno A, Hong SM, Fu B, Lin MT, Calhoun ES, Kamiyama M, Walter K, Nikolskaya T, Nikolsky Y, Hartigan J, Smith DR, Hidalgo M, Leach SD, Klein AP, Jaffee EM, Goggins M, Maitra A, Iacobuzio-Donahue C, Eshleman JR, Kern SE, Hruban RH, Karchin R, Papadopoulos N, Parmigiani G, Vogelstein B, Velculescu VE, Kinzler KW. Core signaling pathways in human pancreatic cancers revealed by global genomic analyses. Science. 2008 Sep 26;321(5897):1801-6. doi: 10.1126/science.1164368. Epub 2008 Sep 4. PMID 18772397
- [Background] Ko AH, Hwang J, Venook AP, Abbruzzese JL, Bergsland EK, Tempero MA. Serum CA19-9 response as a surrogate for clinical outcome in patients receiving fixed-dose rate gemcitabine for advanced pancreatic cancer. Br J Cancer. 2005 Jul 25;93(2):195-9. doi: 10.1038/sj.bjc.6602687. PMID 15999098
- [Background] Nguyen KT, Kalyan A, Beasley HS, Singhi AD, Sun W, Zeh HJ, Normolle D, Bahary N. Gemcitabine/nab-paclitaxel as second-line therapy following FOLFIRINOX in metastatic/advanced pancreatic cancer-retrospective analysis of response. J Gastrointest Oncol. 2017 Jun;8(3):556-565. doi: 10.21037/jgo.2017.01.23. PMID 28736642
- [Background] Maitra A, Hruban RH. Pancreatic cancer. Annu Rev Pathol. 2008;3:157-88. doi: 10.1146/annurev.pathmechdis.3.121806.154305. PMID 18039136
- [Background] Masamune A, Shimosegawa T. Signal transduction in pancreatic stellate cells. J Gastroenterol. 2009;44(4):249-60. doi: 10.1007/s00535-009-0013-2. Epub 2009 Mar 7. PMID 19271115
- [Background] Ponder BA. Cancer genetics. Nature. 2001 May 17;411(6835):336-41. doi: 10.1038/35077207. PMID 11357140
- [Background] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Background] Ueno H, Ioka T, Ikeda M, Ohkawa S, Yanagimoto H, Boku N, Fukutomi A, Sugimori K, Baba H, Yamao K, Shimamura T, Sho M, Kitano M, Cheng AL, Mizumoto K, Chen JS, Furuse J, Funakoshi A, Hatori T, Yamaguchi T, Egawa S, Sato A, Ohashi Y, Okusaka T, Tanaka M. Randomized phase III study of gemcitabine plus S-1, S-1 alone, or gemcitabine alone in patients with locally advanced and metastatic pancreatic cancer in Japan and Taiwan: GEST study. J Clin Oncol. 2013 May 1;31(13):1640-8. doi: 10.1200/JCO.2012.43.3680. Epub 2013 Apr 1. PMID 23547081
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Von Hoff DD, Ramanathan RK, Borad MJ, Laheru DA, Smith LS, Wood TE, Korn RL, Desai N, Trieu V, Iglesias JL, Zhang H, Soon-Shiong P, Shi T, Rajeshkumar NV, Maitra A, Hidalgo M. Gemcitabine plus nab-paclitaxel is an active regimen in patients with advanced pancreatic cancer: a phase I/II trial. J Clin Oncol. 2011 Dec 1;29(34):4548-54. doi: 10.1200/JCO.2011.36.5742. Epub 2011 Oct 3. PMID 21969517
- [Background] Wu J, Liang C, Chen M, Su W. Association between tumor-stroma ratio and prognosis in solid tumor patients: a systematic review and meta-analysis. Oncotarget. 2016 Oct 18;7(42):68954-68965. doi: 10.18632/oncotarget.12135. PMID 27661111
- [Background] Duda DG, Batchelor TT, Willett CG, Jain RK. VEGF-targeted cancer therapy strategies: current progress, hurdles and future prospects. Trends Mol Med. 2007 Jun;13(6):223-30. doi: 10.1016/j.molmed.2007.04.001. Epub 2007 Apr 25. PMID 17462954
- [Background] Grandinetti CA, Goldspiel BR. Sorafenib and sunitinib: novel targeted therapies for renal cell cancer. Pharmacotherapy. 2007 Aug;27(8):1125-44. doi: 10.1592/phco.27.8.1125. PMID 17655513
- [Background] Keating GM, Santoro A. Sorafenib: a review of its use in advanced hepatocellular carcinoma. Drugs. 2009;69(2):223-40. doi: 10.2165/00003495-200969020-00006. PMID 19228077
- [Background] Mross K, Frost A, Steinbild S, Hedbom S, Buchert M, Fasol U, Unger C, Kratzschmar J, Heinig R, Boix O, Christensen O. A phase I dose-escalation study of regorafenib (BAY 73-4506), an inhibitor of oncogenic, angiogenic, and stromal kinases, in patients with advanced solid tumors. Clin Cancer Res. 2012 May 1;18(9):2658-67. doi: 10.1158/1078-0432.CCR-11-1900. Epub 2012 Mar 15. PMID 22421192
- [Background] Sartore-Bianchi A, Zeppellini A, Amatu A, Ricotta R, Bencardino K, Siena S. Regorafenib in metastatic colorectal cancer. Expert Rev Anticancer Ther. 2014 Mar;14(3):255-65. doi: 10.1586/14737140.2014.894887. PMID 24559322
- [Background] Rugo HS, Herbst RS, Liu G, Park JW, Kies MS, Steinfeldt HM, Pithavala YK, Reich SD, Freddo JL, Wilding G. Phase I trial of the oral antiangiogenesis agent AG-013736 in patients with advanced solid tumors: pharmacokinetic and clinical results. J Clin Oncol. 2005 Aug 20;23(24):5474-83. doi: 10.1200/JCO.2005.04.192. Epub 2005 Jul 18. PMID 16027439
- [Background] Sun Q, Zhou J, Zhang Z, Guo M, Liang J, Zhou F, Long J, Zhang W, Yin F, Cai H, Yang H, Zhang W, Gu Y, Ni L, Sai Y, Cui Y, Zhang M, Hong M, Sun J, Yang Z, Qing W, Su W, Ren Y. Discovery of fruquintinib, a potent and highly selective small molecule inhibitor of VEGFR 1, 2, 3 tyrosine kinases for cancer therapy. Cancer Biol Ther. 2014;15(12):1635-45. doi: 10.4161/15384047.2014.964087. PMID 25482937
- [Background] Kuhnz W, Gieschen H. Predicting the oral bioavailability of 19-nortestosterone progestins in vivo from their metabolic stability in human liver microsomal preparations in vitro. Drug Metab Dispos. 1998 Nov;26(11):1120-7. PMID 9806955
- [Background] Obach RS. Prediction of human clearance of twenty-nine drugs from hepatic microsomal intrinsic clearance data: An examination of in vitro half-life approach and nonspecific binding to microsomes. Drug Metab Dispos. 1999 Nov;27(11):1350-9. PMID 10534321
- [Background] Qian H, Fan S, Li K, Sai Y, Su W, Chen Q, Liu Y, Li T, Wang W, Jia J, Yu C, Liu Y. Effects of a High-fat Meal on the Pharmacokinetics of the VEGFR Inhibitor Fruquintinib: A Randomized Phase I Study in Healthy Subjects. Clin Ther. 2019 Aug;41(8):1537-1544. doi: 10.1016/j.clinthera.2019.05.014. Epub 2019 Jul 1. PMID 31272709
- [Background] Cao J, Zhang J, Peng W, Chen Z, Fan S, Su W, Li K, Li J. A Phase I study of safety and pharmacokinetics of fruquintinib, a novel selective inhibitor of vascular endothelial growth factor receptor-1, -2, and -3 tyrosine kinases in Chinese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2016 Aug;78(2):259-69. doi: 10.1007/s00280-016-3069-8. Epub 2016 Jun 14. PMID 27299749
- [Background] Xu RH, Li J, Bai Y, Xu J, Liu T, Shen L, Wang L, Pan H, Cao J, Zhang D, Fan S, Hua Y, Su W. Safety and efficacy of fruquintinib in patients with previously treated metastatic colorectal cancer: a phase Ib study and a randomized double-blind phase II study. J Hematol Oncol. 2017 Jan 19;10(1):22. doi: 10.1186/s13045-016-0384-9. PMID 28103904
- [Background] Li J, Qin S, Xu RH, Shen L, Xu J, Bai Y, Yang L, Deng Y, Chen ZD, Zhong H, Pan H, Guo W, Shu Y, Yuan Y, Zhou J, Xu N, Liu T, Ma D, Wu C, Cheng Y, Chen D, Li W, Sun S, Yu Z, Cao P, Chen H, Wang J, Wang S, Wang H, Fan S, Hua Y, Su W. Effect of Fruquintinib vs Placebo on Overall Survival in Patients With Previously Treated Metastatic Colorectal Cancer: The FRESCO Randomized Clinical Trial. JAMA. 2018 Jun 26;319(24):2486-2496. doi: 10.1001/jama.2018.7855. PMID 29946728
- [Background] Schmidinger M. Understanding and managing toxicities of vascular endothelial growth factor (VEGF) inhibitors. EJC Suppl. 2013 Sep;11(2):172-91. doi: 10.1016/j.ejcsup.2013.07.016. No abstract available. PMID 26217127